CLINICAL TRIAL: NCT03926910
Title: Test of Ventricular Stimulation as Immediate Predictor of Hypovolemia After Cardiac Surgery: Non-randomized Open Label Trial.
Brief Title: Ventricular Stimulation as Predictor of Hypovolemia After Cardiac Surgery
Acronym: TESTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018/13
Record Dates: First submitted 2019-04-17; First posted 2019-04-25 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Cardiac Surgery; Hypovolemia
Keywords: Preload-dependency; hypotension; cardiac surgery; delta PP; PLR; Fluid responsiveness
MeSH Terms: conditions — Hypovolemia; Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VESAP (Experimental): patient receiving stimulation test to detect hypovolemia
  Interventions: Diagnostic Test: Detection of hypovolemia using a ventricular stimulation without atrial pacing

INTERVENTIONS:
Diagnostic Test: Detection of hypovolemia using a ventricular stimulation without atrial pacing — Upon the return in intensive care:
  * Baseline measurements: 1) Three measurements of blood pressure during inspiration and 3 during expiration will be collected for averaging systolic blood pressure, diastolic blood pressure, mean arterial pressure and ΔPP. Data from a pulmonary artery catheter will be also collected.
  * Realization of VESAP pacing with adjustment of the pacemaker (PM) at a heart rate 5 bpm higher than the heart rate of the patient. After 20 seconds of stimulation, recording of the blood pressure curve as done at baseline during at least 3 respiratory cycles,
  * Then vascular filling with 500 ml of physiologic saline solution over 10 minutes and new set of measurement (same than at baseline)
  * Second realization of VESAP pacing, and new set of measurement (same than at Baseline)
  * Then, if the ΔPP is >10%, new vascular filling with 500 ml of physiologic saline solution over 10 min and new set of measurements as previously performed.

SUMMARY:
The purpose of the study is to validate a ventricular pacing test as a predictor of preload dependency in post cardiac surgery patients.

DETAILED DESCRIPTION:
In the immediate postoperative period of cardiac surgery and in intensive care unit (ICU), a systemic arterial hypotension is frequently observed. This hypotension is often due to hypovolemia but also to pump dysfunction and/or vasoplegia. Early recognition of the hypotensive mechanism is necessary because it requires immediate specific treatment.

The interest of a vascular filling is usually estimated by a preload dependence test (fluid responsiveness), showing an increase in the stroke volume when preload is increased according to the Starling the law of the heart. To date, a preload dependency test is usually performed by passive leg raise (PLR) or by measuring the respiratory pulse variation (ΔPP).

The PLR response varies according to the legs venous volume and capacitance. The derivation of ΔPP has been validated in patients intubated, sedated, and ventilated in standard conditions, in sinus rhythm but the ΔPP directly displayed by the monitors is unreliable and the manual calculation on pressure curve is fastidious. Faced with these difficulties, the trend is to realize a blind filling with physiologic saline solution and to judge his interest on clinical and / or hemodynamic criteria.

After cardiac surgery, ventricular epicardial electrodes are systematically placed allowing a temporary stimulation by an external pacemaker in case of postoperative atrio-ventricular blocks. The ventricular stimulation without atrial pacing (VESAP) leads to a loss of the atrial systole and therefore a decrease in the left ventricular preload. During the functional test of epicardial electrodes at a frequency greater than the patient's, it is possible to observe in certain circumstances a decrease of the arterial blood pressure, but of varying importance.

The investigators suspect that the eventual fall in blood pressure during a ventricular pacing test, could be correlated with preload dependence. Therefore, investigator hypothesize that ventricular pacing can be used to realize a functional testing of preload dependence, easy to achieve. Indeed, if doctors admit that during a brief ventricular stimulation, heart rate and systemic vascular resistance remain unchanged, the drop in blood pressure should reflect the decrease in stroke volume.

The main objective of this study is to demonstrate that the response to VESAP can predict the preload dependence of patients after a cardiac surgery. The primary endpoint will study the predictive value of the change in blood pressure during the VESAP and the change in stroke volume after an infusion of 500 cc of crystalloid solution. Secondary endpoints will 1) compare the predictive values of the VESAP and ΔPP; 2) look for pertinent VESAP threshold in correlation with the expected increase in stroke volume; and 3) collection of the possible complications due to the VESAP.

30 patients will be enrolled in this monocentric, open label, non-randomized study.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old,
* Programmed for cardiac surgery with the need for invasive hemodynamic monitoring (pulmonary artery catheter) according to the recommendations:

  * Euroscore with predicted mortality> 10%
  * Left ventricular ejection fraction (LVEF) <40%
  * Left ventricular ejection fraction (LVEF) <50% for mitral insufficiency
  * pulmonary artery hypertension (PAH)> 50 mmHg
  * Tricuspid insufficiency> 3.4 m / s
  * Tricuspid annular plane systolic excursion (TAPSE) <16 mm
  * Dilatation of the inferior vena cava under respiratory collapse
* Sinus rhythm in immediate postoperative period,
* Sedated with mechanical ventilation,
* Having given their written participation consent in accordance with the regulations,
* Benefiting from a social security

Exclusion Criteria:

* Pregnant or lactating women,
* Patient under guardianship, Under curatorship or court of justice,
* Discomfort to communication or neuropsychic disorders,Inability to understand, to read or to write the French language,
* Patients for whom a fluids overload seems obvious to the intensivist and for whom a crystalloids filling would be contraindicated,
* Patients for whom respiratory changes in pulse pressure (ΔPP) measurement is not validated: patients with spontaneous ventilation, atrial fibrillation, non-sedated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2020-10-13 (Actual); Study Completion 2020-10-14 (Actual)

PRIMARY OUTCOMES:
Evaluate the correlation between thes stimulation test and the cardiac output | 1 hour
  Measure the cardiac flow before and after the VESAP, and after an infusion of 500 cc of crystalloid solution.

SECONDARY OUTCOMES:
Collection of the possible complications due to the VESAP | 2 hours and 24 hours
  Number of participants with low blood presseur or with heart rhythm disorder.
Evaluate the correlation between the VESAP and the ΔP | 1 hour
  Measure the of the blood presser before and after stimulation test and after an infusion of 500 cc of crystalloid solution
Look for pertinent VESAP threshold in correlation with the expected increase in stroke volume | 1 hour
  Measure the of the strocke volume before and after stimulation test and after an infusion of 500 cc of crystalloid solution

CONTACTS AND LOCATIONS:
Overall Officials: Philippe ESTAGNASIÉ, MD, Principal Investigator — CMC Ambroise Paré
Locations (1):
- CMC Ambroise Paré, Neuilly-sur-Seine, Neuilly Sur Seine Ile de France, France